CLINICAL TRIAL: NCT06474273
Title: A Multicenter Randomized Controlled Trial to Treat Acute t Cell Mediated Rejection in Kidney and Kidney-pancreas Transplant Recipients
Brief Title: TACKLE-IT Trial - Treat Acute T Cell Rejection With Evidence and Confidence in Kidney Transplant Recipients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sydney (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWCT051274
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Rejection; Transplant, Kidney; Rejection; Transplant, Pancreas
Keywords: Acute T cell mediated rejection
MeSH Terms: conditions — Rejection, Psychology | interventions — Methylprednisolone; Prednisone

STUDY DESIGN:
Intervention Model Description: 2x2 factorial, triple-blind, non-inferiority, RCT of lower vs higher dose IV MP (methylprednisolone), and lower vs higher oral prednisone dose augmentation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: As a triple-blind study, all investigators, research staff, clinicians, outcome assessors, data analysts and participants will be blinded to the allocation of the IV MP treatment comparisons.
  All key stakeholders including the global steering committee, the site investigators, and the trial management committee (TMC) will remain blinded to the individual patient randomization and the aggregate data that may reveal the unblinded outcomes. All researchers responsible for the analysis will remain blinded for the duration of the trial. Only the members of the Data Safety Monitoring Board (DSMB) and the independent statistician supporting their work will be unblinded prior to study completion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Lower dose IV methylprednisolone x Lower dose oral prednisone (Experimental): Lower dose IV MP (250 mg daily x 3 days in adults or 150 mg/m² daily x 3, or to a max 250 mg/dose in children (<18 years), with lower dose (25mg daily x 7 days, or 15mg/m² for those < 18 years ) oral prednisone augmentation then return to standard prednisone.
  Interventions: Drug: Methylprednisolone; Drug: Prednisone
- Lower dose IV methylprednisolone x Higher dose oral prednisone (Experimental): Lower dose IV MP (250 mg daily x 3 in adults or 150 mg/m² daily x 3, or to a max 250 mg/dose in children (<18 years), with higher dose (50mg daily x 7 , or 30mg/m² daily x 7 for those < 18 years) oral prednisone augmentation then return to standard prednisone.
  Interventions: Drug: Methylprednisolone; Drug: Prednisone
- Higher dose IV methylprednisolone x lower dose oral prednisone (Active Comparator): Higher dose IV MP (500mg daily x 3 in adults or 300 mg/m² daily x 3 or to a max 500 mg/dose in children (<18 years), with lower dose (25mg daily x 7 days, or 15mg/m² for those < 18 years) oral prednisone augmentation then return to standard prednisone.
  Interventions: Drug: Methylprednisolone; Drug: Prednisone
- Higher dose IV methylprednisolone x higher dose oral prednisone (Active Comparator): Higher dose IV MP (500 mg daily x 3 in adults or 300 mg/m² daily x 3 or to a max 500 mg/dose in children (<18 years), with higher dose (50mg daily x 7 days, or 30mg/m² for those < 18 years) oral prednisone augmentation, then return to standard prednisone.
  Interventions: Drug: Methylprednisolone; Drug: Prednisone

INTERVENTIONS:
Drug: Methylprednisolone — IV Methylprednisolone
  Other Names: IV MP
Drug: Prednisone — Oral prednisone augmentation

SUMMARY:
After a kidney or a simultaneous kidney-pancreas transplant, some patients may face problems with their new organs. This happens because the body sometimes makes a mistake and tries to get rid of the organ. This problem is called rejection. One type of rejection is known as Acute T cell mediated rejection (TCMR). This can lead to many problems or even stop the transplant from working.

Doctors give strong steroids to treat this problem, but there are no rules for how much steroid to give. Too much steroids can cause problems like heart and bone problems, bad infections, and weight gain. That is why we need to find the right dose of steroids for each person to treat this.

TACKLE-IT is a study that will try to find the right steroid dose for treating rejection.

DETAILED DESCRIPTION:
TACKLE-IT is an international, multi-centre, 2x2 factorial, triple-blind, non-inferiority registry-embedded, randomised controlled trial (RCT) that compares the effectiveness and safety of high vs low dose IV MP, and high vs low dose oral prednisone taper as the first-line therapy for acute TCMR in kidney and SPK transplant recipients. This RCT was conceived and developed through extensive consultation and collaboration with our key stakeholders, including transplant recipients with lived experience and the International TCMR Working Group with sponsorship by 4 international transplant societies (The Transplantation Society (TTS), American Society of Transplantation (AST), European Society of Transplantation (ESOT) and Transplant Society of Australia and New Zealand (TSANZ). TACKLE-IT is led by an international multi-disciplinary team of transplant health professionals, clinical trialists, biostatisticians, health economist, social scientist, consumers.

TACKLE-IT will address the critical unmet need and resolve a decades-long unanswered question, 'What is the minimally acceptable, safe and effective steroid dose for the treatment of acute TCMR in kidney and SPK transplant recipients?'

ELIGIBILITY:
Inclusion Criteria:

* Participants or their legal guardian must be able to understand and provide written informed consent;
* Stated willingness to comply with all study procedures and availability for the duration of the study;
* All ethnic and gender groups will have equal access to the study;
* All children (aged 2+ years) and adults who have received a kidney or SPK transplant with biopsy proven acute TCMR (≥ Banff borderline (minimum i1 score) whether clinical or subclinical).

Exclusion Criteria:

* Mixed rejection.
* Active or chronic active ABMR.
* Chronic active TCMR. *Patients with concomitant acute TCMR and chronic active TCMR will not be excluded from the trial.
* Isolated v1 without inflammation.
* Concurrent renal disease, such as recurrent glomerulonephritis or polyomavirus nephropathy.
* Active malignancies or active infection that preclude immunosuppression augmentation.
* Use of other immunomodulatory agents, including, but not limited to, Rituximab, Anti-TNF monoclonal antibody, Belatacept, Abatacept, Janus kinase inhibitors, Eculizumab, Pegcetacoplan.
* Enrolment in other interventional drug trials.
* Use of other investigational agents.
* Unable to adhere to the study protocol.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Histological resolution of biopsy-proven acute rejection | 12 weeks post-randomization
  Histological resolution of biopsy-proven acute rejection is defined by the absence of any biopsy-proven acute rejection (BPAR) on follow-up biopsy, including <Banff Borderline (i1 t1), mixed rejection, ABMR and chronic active TCMR using Banff 2022 criteria.
Improvement in allograft function | 12 weeks post-randomization
  Baseline serum creatinine is defined by an average of three serum creatinine measures: i) first serum creatinine preceding randomisation , ii) serum creatinine at the time of randomisation, iii) serum creatinine at the time of the first IV MP.
  Reduction in serum creatinine ≥20% is defined as the relative reduction in serum creatinine from baseline and at 12 weeks after randomisation.
Avoidance of rescue therapies within 12 weeks post-randomization to achieve histological resolution and/or improvement in allograft function | 12 weeks post-randomization
  Use of rescue therapy is defined as: the use of any adjunctive T and B cell depleting therapies such as intravenous thymoglobulin, alemtuzumab, bortezomib, or rituximab, or additional doses of IV MP within the first 12 weeks after randomization.

SECONDARY OUTCOMES:
Estimated glomerular filtration rate (eGFR) | At 12, 24 and 48 weeks post-randomization
  * Absolute eGFR (2021 CKD-EPI eGFR without race modifier for adults, and the CKiD U25 equation to estimate GFR in children &amp;amp;amp;amp;amp;lt; 18 years) 12, 24 and 48 weeks.
  * Decline in eGFR (slope) from randomization to 48 weeks.
All cause death and death-censored graft loss | At 12 weeks post-randomization
  All cause death and death-censored graft loss have been identified as the core outcomes for kidney transplant recipients. However, death and death-censored graft loss are anticipated to have a very low incidence at the 12 weeks post-randomization primary outcome ascertainment and were therefore not included in the primary composite outcome. They will be reported as principal secondary endpoints.
Urine albumin: creatinine ratios | At 12, 24 and 48 weeks post-randomization
  Urine ACR is measured as standard of care. Rationale: ACR screens for graft dysfunction and is a marker for graft outcomes
Quality of life (QoL) | Baseline (at randomization), 12 weeks , 24 weeks , and 48 weeks post-randomization
  QoL will be assessed using the EuroQol-5 Dimension-5 Level (EQ-5D-5L) for adult participants (aged ≥18 years). For paediatric participants (aged 2-17 years), age-appropriate versions of the EuroQol Youth version (EQ-5D-Y) will be used as follows:
  * Ages 4-7: EQ-5D-Y proxy version
  * Ages 8-11: EQ-5D-Y self-report version
  * Ages 12-15: EQ-5D-Y self-report version
  * Age ≥16: EQ-5D-5L adult version
  Both the EQ-5D-5L and EQ-5D-Y report utility scores ranging from -0.281 to 1 (EQ-5D-5L UK value set) and -0.109 to 1 (EQ-5D-Y, proxy or self-report), where 1 represents perfect health, 0 represents a health state equivalent to death, and negative scores represent health states worse than death. Higher scores indicate better health-related quality of life.
Cancer | Anytime from randomization to 48 weeks
  All types and sites
Trajectories of serum creatinine changes | From randomization to 48 weeks post-randomization
  An average of three serum creatinine measures will be considered as baseline serum creatinine measures: i) first serum creatinine preceding randomization, ii) serum creatinine at the time of randomisation, iii) serum creatinine at the time of the first IV MP.
Development of acute antibody mediated rejection (ABMR) and mixed rejection (concomitant ABMR + TCMR) | 48 weeks post-randomization
  ABMR and mixed rejection are defined according to the Banff 2022 criteria
Infections (including those requiring antimicrobials and hospitalisation) | Anytime from randomization to 48 weeks post-randomization
  All types and number of events related to infections that required antimicrobials and hospitalisation for infections will be recorded.
Development of chronic fibrosis in the allograft | Baseline to 12 weeks post-randomization
  This is defined as a change in ci and ct scores (a marker of interstitial fibrosis and tubular atrophy, measurement of fibrosis, defined by the Banff 2022 criteria)

OTHER OUTCOMES:
Steroid-related adverse effects | 3 days post randomisation, 7 days post randomisation, week 12 post-randomisation, week 24 post-randomisation and week 48 post-randomisation
  Adaption from the Steroid Patient Reported Outcome (Steroid PRO).
Integrative Box Risk Prediction Score (iBOX) | Week 13 to week 48 post-randomisation
  Graft survival prediction will be assessed using the Integrative Box Risk Prediction Score (iBOX), a validated composite risk prediction tool for kidney transplant outcomes. The iBOX score integrates clinical, functional, and immunological parameters including serum creatinine, proteinuria, biopsy findings, and presence of donor-specific antibodies to estimate the risk of allograft failure. The iBox score essentially assigns a numerical value based on these parameters, indicating the risk of allograft loss (kidney transplant failure).
Economic evaluation: Incremental costs and benefits | During the 52-week follow up period
  Economic evaluation to compare the incremental benefits (in QALYs) and costs between the treatment arms.
Process evaluation: patients' and clinicians' perspectives on the treatment of acute TCMR | Anytime between week 12 and 48 of the trial
  Semi-structured interviews will be conducted to elicit patients' perspectives and experiences of having acute TCMR, the adverse effects of the treatments. Health professionals' will also be interviewed to elicit their perspectives and experiences regarding the barriers, challenges, and enablers for implementing the intervention, the perceived benefits, and harms of the intervention and how the intervention should be delivered such that maximal interactions of the intervention are reached for the intended participants.
T cell receptor repertoire | Week 13 to week 48 post-randomization
  To characterise and compare the T cell receptor (TCR) repertoire in transplant recipients who were responsive and not responsive to the various corticosteroid dosing strategies in acute TCMR.
Life participation | Randomisation, week 12 post-randomization, week 24 post-randomization and week 48 post-randomization
  Life participation will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS®) Ability to Participate in Social Roles and Activities - Short Form 4a (SF4a). This instrument measures perceived ability to perform usual social roles and activities.
  Scores are reported as T-scores standardized to the general U.S. population (mean = 50, SD = 10).
  * Minimum score: 20
  * Maximum score: 80
  Higher scores indicate better ability to participate in social roles and activities (i.e., a more favorable outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Germaine Wong, PhD, FRACP, Principal Investigator — University of Sydney; Julie Ho, FRCPC, Principal Investigator — University of Manitoba
Locations (25):
- Australia (11):
  - John Hunter Hospital, Lambton, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - The Sydney Children's Hospital Network, Westmead, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Royal Perth Children's hospital, Nedlands, Western Australia
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
- Canada (13):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Transplant Manitoba, adult, Winnipeg, Manitoba
  - Transplant Manitoba, pediatric, Winnipeg, Manitoba
  - Dalhousie University, Halifax, Nova Scotia
  - Western University, London, Ontario
  - University of Toronto - St Michael Hospital, Toronto, Ontario
  - University of Toronto - Hospital for Sick Kids, Toronto, Ontario
  - University of Toronto, Toronto, Ontario
  - McGill University, Montreal, Quebec
  - University of Montreal, Montreal, Quebec
  - University of Laval, Québec, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan
- Auckland City Hospital, Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
The data collected for the study, including individual patient data and a data dictionary that defines each field in the data set, will be made available as deidentified participant data to researchers who propose to use the data for individual patient data meta-analysis. Data will be shared following approval of the proposal by the corresponding author and a signed data access agreement, beginning 2 years following main publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study protocol, SAP, ICF will be provided 3 months after registration. The Clinical study report and code will be provided after completion of the trial.
Access Criteria: All IPD data arising from the trial will be shared 2 years after publication of the main results.

REFERENCES:
- [Background] Wiebe C, Gibson IW, Blydt-Hansen TD, Karpinski M, Ho J, Storsley LJ, Goldberg A, Birk PE, Rush DN, Nickerson PW. Evolution and clinical pathologic correlations of de novo donor-specific HLA antibody post kidney transplant. Am J Transplant. 2012 May;12(5):1157-67. doi: 10.1111/j.1600-6143.2012.04013.x. Epub 2012 Mar 19. PMID 22429309
- [Background] Wiebe C, Kosmoliaptsis V, Pochinco D, Gibson IW, Ho J, Birk PE, Goldberg A, Karpinski M, Shaw J, Rush DN, Nickerson PW. HLA-DR/DQ molecular mismatch: A prognostic biomarker for primary alloimmunity. Am J Transplant. 2019 Jun;19(6):1708-1719. doi: 10.1111/ajt.15177. Epub 2018 Dec 15. PMID 30414349
- [Background] Wiebe C, Rush DN, Gibson IW, Pochinco D, Birk PE, Goldberg A, Blydt-Hansen T, Karpinski M, Shaw J, Ho J, Nickerson PW. Evidence for the alloimmune basis and prognostic significance of Borderline T cell-mediated rejection. Am J Transplant. 2020 Sep;20(9):2499-2508. doi: 10.1111/ajt.15860. Epub 2020 Apr 9. PMID 32185878
- [Background] Nickerson PW, Balshaw R, Wiebe C, Ho J, Gibson IW, Bridges ND, Rush DN, Heeger PS. A noninferiority design for a delayed calcineurin inhibitor substitution trial in kidney transplantation. Am J Transplant. 2021 Apr;21(4):1503-1512. doi: 10.1111/ajt.16311. Epub 2020 Oct 6. PMID 32956576
- [Background] Rampersad C, Balshaw R, Gibson IW, Ho J, Shaw J, Karpinski M, Goldberg A, Birk P, Rush DN, Nickerson PW, Wiebe C. The negative impact of T cell-mediated rejection on renal allograft survival in the modern era. Am J Transplant. 2022 Mar;22(3):761-771. doi: 10.1111/ajt.16883. Epub 2021 Nov 24. PMID 34717048
- [Background] Ho J, Okoli GN, Rabbani R, Lam OLT, Reddy VK, Askin N, Rampersad C, Trachtenberg A, Wiebe C, Nickerson P, Abou-Setta AM. Effectiveness of T cell-mediated rejection therapy: A systematic review and meta-analysis. Am J Transplant. 2022 Mar;22(3):772-785. doi: 10.1111/ajt.16907. Epub 2021 Dec 10. PMID 34860468
- [Background] Nankivell BJ, Shingde M, Keung KL, Fung CL, Borrows RJ, O'Connell PJ, Chapman JR. The causes, significance and consequences of inflammatory fibrosis in kidney transplantation: The Banff i-IFTA lesion. Am J Transplant. 2018 Feb;18(2):364-376. doi: 10.1111/ajt.14609. Epub 2018 Jan 3. PMID 29194971
- [Background] Tong A, Budde K, Gill J, Josephson MA, Marson L, Pruett TL, Reese PP, Rosenbloom D, Rostaing L, Warrens AN, Wong G, Craig JC, Crowe S, Harris T, Hemmelgarn B, Manns B, Tugwell P, Van Biesen W, Wheeler DC, Winkelmayer WC, Evangelidis N, Sautenet B, Howell M, Chapman JR. Standardized Outcomes in Nephrology-Transplantation: A Global Initiative to Develop a Core Outcome Set for Trials in Kidney Transplantation. Transplant Direct. 2016 May 19;2(6):e79. doi: 10.1097/TXD.0000000000000593. eCollection 2016 Jun. PMID 27500269
- [Background] Sautenet B, Tong A, Chapman JR, Warrens AN, Rosenbloom D, Wong G, Gill J, Budde K, Rostaing L, Marson L, Josephson MA, Reese PP, Pruett TL, Evangelidis N, Craig JC. Range and Consistency of Outcomes Reported in Randomized Trials Conducted in Kidney Transplant Recipients: A Systematic Review. Transplantation. 2018 Dec;102(12):2065-2071. doi: 10.1097/TP.0000000000002278. PMID 29781954
- [Background] Sautenet B, Tong A, Manera KE, Chapman JR, Warrens AN, Rosenbloom D, Wong G, Gill J, Budde K, Rostaing L, Marson L, Josephson MA, Reese PP, Pruett TL, Hanson CS, O'Donoghue D, Tam-Tham H, Halimi JM, Shen JI, Kanellis J, Scandling JD, Howard K, Howell M, Cross N, Evangelidis N, Masson P, Oberbauer R, Fung S, Jesudason S, Knight S, Mandayam S, McDonald SP, Chadban S, Rajan T, Craig JC. Developing Consensus-Based Priority Outcome Domains for Trials in Kidney Transplantation: A Multinational Delphi Survey With Patients, Caregivers, and Health Professionals. Transplantation. 2017 Aug;101(8):1875-1886. doi: 10.1097/TP.0000000000001776. PMID 28738403
- [Background] Tong A, Gill J, Budde K, Marson L, Reese PP, Rosenbloom D, Rostaing L, Wong G, Josephson MA, Pruett TL, Warrens AN, Craig JC, Sautenet B, Evangelidis N, Ralph AF, Hanson CS, Shen JI, Howard K, Meyer K, Perrone RD, Weiner DE, Fung S, Ma MKM, Rose C, Ryan J, Chen LX, Howell M, Larkins N, Kim S, Thangaraju S, Ju A, Chapman JR; SONG-Tx Investigators. Toward Establishing Core Outcome Domains For Trials in Kidney Transplantation: Report of the Standardized Outcomes in Nephrology-Kidney Transplantation Consensus Workshops. Transplantation. 2017 Aug;101(8):1887-1896. doi: 10.1097/TP.0000000000001774. PMID 28737661
- [Background] Tong A, Sautenet B, Poggio ED, Lentine KL, Oberbauer R, Mannon R, Murphy B, Padilla B, Chow KM, Marson L, Chadban S, Craig JC, Ju A, Manera KE, Hanson CS, Josephson MA, Knoll G; SONG-Tx Graft Health Workshop Investigators. Establishing a Core Outcome Measure for Graft Health: A Standardized Outcomes in Nephrology-Kidney Transplantation (SONG-Tx) Consensus Workshop Report. Transplantation. 2018 Aug;102(8):1358-1366. doi: 10.1097/TP.0000000000002125. PMID 29470347
- [Background] Ju A, Josephson MA, Butt Z, Jowsey-Gregoire S, Tan J, Taylor Q, Fowler K, Dobbels F, Caskey F, Jha V, Locke J, Knoll G, Ahn C, Hanson CS, Sautenet B, Manera K, Craig JC, Howell M, Rutherford C, Tong A, Harden P, Hawley C, Holdaas H, Israni A, Jesse M, Kane B, Kanellis J, Kiberd B, Kim J, Larsen C, Leichtman A, Lentine K, Malone A, Mannon R, Oberbauer R, Patzer R, Peipert JD, Phan HA, Poggio E, Reed R, Scandling J, Tang I, Watson C, Contrares D, Contreras P, Cross D, Juodvalkis E, Koide D, Koide J, Kozarewicz A, Kozarewicz L, Kozarewicz R, Koritala A, Lisiecki E, Lipuma C, Lyman M, Mueller R, Mueller G, Noble L, Nolan N, Nolan S, Thomas J, Urbancyzk L, Zerante J, Zerante S; SONG-Tx Life Participation Workshop Investigators; Health professionals (*includes 2 patients from the SONG-Tx Graft Health Expert Working Group); Patients and family members. Establishing a Core Outcome Measure for Life Participation: A Standardized Outcomes in Nephrology-kidney Transplantation Consensus Workshop Report. Transplantation. 2019 Jun;103(6):1199-1205. doi: 10.1097/TP.0000000000002476. PMID 30300284
- [Background] Ju A, Chow BY, Ralph AF, Howell M, Josephson MA, Ahn C, Butt Z, Dobbels F, Fowler K, Jowsey-Gregoire S, Jha V, Locke JE, Tan JC, Taylor Q, Rutherford C, Craig JC, Tong A. Patient-reported outcome measures for life participation in kidney transplantation: A systematic review. Am J Transplant. 2019 Aug;19(8):2306-2317. doi: 10.1111/ajt.15267. Epub 2019 Feb 28. PMID 30664327